CLINICAL TRIAL: NCT03837470
Title: Evaluation of Renal Sodium Excretion After Salt Loading in Heart Failure With Preserved Ejection Fraction
Acronym: ERES-HFpEF
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Adhish Agarwal (Other)
Collaborators: University of Utah Center for Clinical and Translational Science (Unknown)
Responsible Party: Sponsor-Investigator, Adhish Agarwal, Associate Professor, Nephrology, University of Utah
Organization: University of Utah (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB_00112270
Record Dates: First submitted 2019-02-08; First posted 2019-02-12 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Heart Failure With Preserved Ejection Fraction
MeSH Terms: interventions — Sodium Chloride; Saline Solution; Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Saline Loading and Diuretic Challenge (Experimental): Subjects receive intravenous infusion of 0.9% Sodium Chloride, followed by diuretic challenge with bolus injection of Furosemide 40 mg
  Interventions: Drug: 0.9% Sodium Chloride; Drug: Furosemide 40 mg

INTERVENTIONS:
Drug: 0.9% Sodium Chloride — Intravenous infusion of 0.25ml/kg/min of 0.9% sodium chloride intravenously for a total of 60 minutes
  Other Names: normal saline
Drug: Furosemide 40 mg — Bolus intravenous injection of 40 mg furosemide

SUMMARY:
Heart failure (HF) affects 2-3% of the population, and is characterized by impaired sodium balance which results in fluid overload. Ejection fraction, a measure of systolic function, is reduced in only about half of all HF patients. Incidence of heart failure with preserved ejection fraction (HFpEF) has increased in the last 20 years making it a growing public health problem. Currently, most patients admitted to the hospital with heart failure have preserved rather than reduced ejection fractions. However, to date it remains unknown why patients with HFpEF retain salt and water. The hypothesis is that patients with clinical HFpEF have an impaired renal response to salt loading, intravascular expansion and diuretics. Characterization of the salt and water excretory renal response to intravascular salt, fluid and diuretic load in patients with HFpEF will provide insight into the pathophysiology of HFpEF, and may help in the development of novel strategies to target renal sodium handling in patients with HFpEF. This characterization is the primary objective of this pilot project.

DETAILED DESCRIPTION:
In patients with heart failure with reduced ejection fraction (HFrEF), poor renal perfusion and neuro-hormonal activation cause renal salt and water retention. In contrast to HFrEF, patients with HFpEF have blunted neuro-hormonal activation, and other mechanisms likely cause fluid overload. Investigators have proposed several mechanisms including inflammatory state, endothelial dysfunction, decreased vascular compliance, pulmonary hypertension, and reduced nitric oxide (NO) bioavailability. However, the etiology and pathophysiology of fluid overload in HFpEF patients remains controversial.

Renal dysfunction is common in patients with HFpEF, and is associated with cardiac remodeling. HFpEF is associated with coronary microvascular endothelial activation and oxidative stress, which through reduction of NO dependent signaling contributes to the high cardiomyocyte stiffness and hypertrophy. Plasma sodium stiffens vascular endothelium and reduces NO release. Thus, renal sodium retention may play a pivotal role in the pathophysiology of HFpEF. Patients with HFrEF indeed have abnormal renal sodium excretion in response to salt load; however, it remains unclear if patients with HFpEF also have an impaired renal sodium excretion in response to a salt load, volume expansion or diuretics.

Since (as noted above) renal sodium retention may play an important role in the pathophysiology of HFpEF, it may be critically important to characterize renal sodium handling in patients with clinical HFpEF in response to salt loading, intravascular expansion and diuretic challenge. Impaired sodium excretion has been previously demonstrated in response to volume expansion in pre-clinical systolic and diastolic dysfunction, but not in patients with clinical HFpEF. Further, it is of note that this impairment in renal sodium excretion is rescued by exogenous B-type natriuretic peptide (BNP), which is a natriuretic peptide that is increased in most patients with HFpEF. It is possible, although not reported, that baseline BNP [which is commonly assessed by N-terminal prohormone of BNP (NT-proBNP)] levels affect renal sodium handling in HFpEF patients in response to salt and volume load, or diuretic challenge. It is also unknown if baseline kidney function, measured by estimated glomerular filtration rate (eGFR), affects natriuresis in patients with HFpEF after salt loading or diuretic challenge. Renal tubular function may also have important effects on salt retention in HF patients.

Characterization of the natriuretic response to intravascular salt and volume load and diuretic challenge, and of tubular function, in patients with HFpEF will provide insight into the pathophysiology of HFpEF, and may help in the development of novel strategies to target renal sodium handling in patients with HFpEF.

ELIGIBILITY:
Inclusion Criteria:

* History of chronic (> 6 months) heart failure with current New York Heart Association II-III symptoms
* Left ventricular ejection fraction > 50% on a clinically indicated echocardiogram obtained within last 12 months
* Clinical compensated heart failure
* On constant medical therapy for heart failure; without changes in heart failure medication regimen (including diuretics) for previous 14 days and not expected to change in the next 2 days

Exclusion Criteria:

* Unable to comply with protocol or procedures
* Uncontrolled severe hypertension: systolic blood pressure > 160 mmHg
* Significant renal impairment as defined by estimated glomerular filtration rate < 30ml/min/1.73m^2 determined by Chronic Kidney Disease - Epidemiology Collaboration equation
* Significant proteinuria (> 0.5 g protein/daily protein or equivalent)
* Body Mass Index > 40 kg/m^2
* Acute coronary syndrome within last 4 weeks
* Coronary revascularization procedures (percutaneous coronary intervention or cardiac artery bypass graft) or valve surgery within 30 days of screening
* Cardiac resynchronization therapy, with or without implantable cardioverter defibrillator within 90 days of screening
* Clinically relevant cardiac valvular disease
* Hypertrophic or restrictive cardiomyopathy, constrictive pericarditis, active myocarditis, active endocarditis, or complex congenital heart disease
* Cirrhosis of the liver
* History of known hydronephrosis
* History of adrenal insufficiency

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Urinary Sodium Excretion | 5 Hours
  Amount of sodium excretion following saline loading and diuretic challenge will be compared between HFpEF patients and controls
Urine Volume | 5 Hours
  Volume of urine collected following saline loading and diuretic challenge will be compared between HFpEF patients and controls

SECONDARY OUTCOMES:
Change in NT-proBNP | 5 Hours
  Average change in NT-proBNP values before and after saline loading and diuretic challenge will be compared between HFpEF patients and controls
Serum Aldosterone | 5 Hours
  Serum Aldosterone levels at baseline, after saline loading and after furosemide administration compared between HFpEF patients and controls
Plasma Renin Activity | 5 Hours
  Plasma renin activity levels at baseline, after saline loading and after furosemide administration compared between HFpEF patients and controls
Plasma Nor-epinephrine | 5 Hours
  Plasma nor-epinephrine levels at baseline, after saline loading and after furosemide administration compared between HFpEF patients and controls

OTHER OUTCOMES:
Urinary Exosomes | 5 Hours
  Sodium transporters in Urinary exosomes will be characterized and compared between HFpEF patients and controls

CONTACTS AND LOCATIONS:
Overall Officials: Adhish Agarwal, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Metra M, Teerlink JR. Heart failure. Lancet. 2017 Oct 28;390(10106):1981-1995. doi: 10.1016/S0140-6736(17)31071-1. Epub 2017 Apr 28. PMID 28460827
- [Background] Dunlay SM, Roger VL, Redfield MM. Epidemiology of heart failure with preserved ejection fraction. Nat Rev Cardiol. 2017 Oct;14(10):591-602. doi: 10.1038/nrcardio.2017.65. Epub 2017 May 11. PMID 28492288
- [Background] Owan TE, Hodge DO, Herges RM, Jacobsen SJ, Roger VL, Redfield MM. Trends in prevalence and outcome of heart failure with preserved ejection fraction. N Engl J Med. 2006 Jul 20;355(3):251-9. doi: 10.1056/NEJMoa052256. PMID 16855265
- [Background] Braunwald E. Heart failure. JACC Heart Fail. 2013 Feb;1(1):1-20. doi: 10.1016/j.jchf.2012.10.002. Epub 2013 Feb 4. PMID 24621794
- [Background] Shah AM, Mann DL. In search of new therapeutic targets and strategies for heart failure: recent advances in basic science. Lancet. 2011 Aug 20;378(9792):704-12. doi: 10.1016/S0140-6736(11)60894-5. PMID 21856484
- [Background] Kitzman DW, Little WC, Brubaker PH, Anderson RT, Hundley WG, Marburger CT, Brosnihan B, Morgan TM, Stewart KP. Pathophysiological characterization of isolated diastolic heart failure in comparison to systolic heart failure. JAMA. 2002 Nov 6;288(17):2144-50. doi: 10.1001/jama.288.17.2144. PMID 12413374
- [Background] Paulus WJ, Tschope C. A novel paradigm for heart failure with preserved ejection fraction: comorbidities drive myocardial dysfunction and remodeling through coronary microvascular endothelial inflammation. J Am Coll Cardiol. 2013 Jul 23;62(4):263-71. doi: 10.1016/j.jacc.2013.02.092. Epub 2013 May 15. PMID 23684677
- [Background] Ter Maaten JM, Damman K, Verhaar MC, Paulus WJ, Duncker DJ, Cheng C, van Heerebeek L, Hillege HL, Lam CS, Navis G, Voors AA. Connecting heart failure with preserved ejection fraction and renal dysfunction: the role of endothelial dysfunction and inflammation. Eur J Heart Fail. 2016 Jun;18(6):588-98. doi: 10.1002/ejhf.497. Epub 2016 Feb 10. PMID 26861140
- [Background] Lam CS, Brutsaert DL. Endothelial dysfunction: a pathophysiologic factor in heart failure with preserved ejection fraction. J Am Coll Cardiol. 2012 Oct 30;60(18):1787-9. doi: 10.1016/j.jacc.2012.08.004. Epub 2012 Oct 3. No abstract available. PMID 23040569
- [Background] Kawaguchi M, Hay I, Fetics B, Kass DA. Combined ventricular systolic and arterial stiffening in patients with heart failure and preserved ejection fraction: implications for systolic and diastolic reserve limitations. Circulation. 2003 Feb 11;107(5):714-20. doi: 10.1161/01.cir.0000048123.22359.a0. PMID 12578874
- [Background] Lam CS, Roger VL, Rodeheffer RJ, Borlaug BA, Enders FT, Redfield MM. Pulmonary hypertension in heart failure with preserved ejection fraction: a community-based study. J Am Coll Cardiol. 2009 Mar 31;53(13):1119-26. doi: 10.1016/j.jacc.2008.11.051. PMID 19324256
- [Background] Takimoto E, Champion HC, Li M, Belardi D, Ren S, Rodriguez ER, Bedja D, Gabrielson KL, Wang Y, Kass DA. Chronic inhibition of cyclic GMP phosphodiesterase 5A prevents and reverses cardiac hypertrophy. Nat Med. 2005 Feb;11(2):214-22. doi: 10.1038/nm1175. Epub 2005 Jan 23. PMID 15665834
- [Background] Zamani P, French B, Brandimarto JA, Doulias PT, Javaheri A, Chirinos JA, Margulies KB, Townsend RR, Sweitzer NK, Fang JC, Ischiropoulos H, Cappola TP. Effect of Heart Failure With Preserved Ejection Fraction on Nitric Oxide Metabolites. Am J Cardiol. 2016 Dec 15;118(12):1855-1860. doi: 10.1016/j.amjcard.2016.08.077. Epub 2016 Sep 15. PMID 27742422
- [Background] Franssen C, Chen S, Unger A, Korkmaz HI, De Keulenaer GW, Tschope C, Leite-Moreira AF, Musters R, Niessen HW, Linke WA, Paulus WJ, Hamdani N. Myocardial Microvascular Inflammatory Endothelial Activation in Heart Failure With Preserved Ejection Fraction. JACC Heart Fail. 2016 Apr;4(4):312-24. doi: 10.1016/j.jchf.2015.10.007. Epub 2015 Dec 9. PMID 26682792
- [Background] Oghlakian GO, Sipahi I, Fang JC. Treatment of heart failure with preserved ejection fraction: have we been pursuing the wrong paradigm? Mayo Clin Proc. 2011 Jun;86(6):531-9. doi: 10.4065/mcp.2010.0841. Epub 2011 May 16. PMID 21576513
- [Background] Gladden JD, Chaanine AH, Redfield MM. Heart Failure with Preserved Ejection Fraction. Annu Rev Med. 2018 Jan 29;69:65-79. doi: 10.1146/annurev-med-041316-090654. PMID 29414252
- [Background] Tschope C, Van Linthout S, Kherad B. Heart Failure with Preserved Ejection Fraction and Future Pharmacological Strategies: a Glance in the Crystal Ball. Curr Cardiol Rep. 2017 Aug;19(8):70. doi: 10.1007/s11886-017-0874-6. PMID 28656481
- [Background] Gori M, Senni M, Gupta DK, Charytan DM, Kraigher-Krainer E, Pieske B, Claggett B, Shah AM, Santos AB, Zile MR, Voors AA, McMurray JJ, Packer M, Bransford T, Lefkowitz M, Solomon SD; PARAMOUNT Investigators. Association between renal function and cardiovascular structure and function in heart failure with preserved ejection fraction. Eur Heart J. 2014 Dec 21;35(48):3442-51. doi: 10.1093/eurheartj/ehu254. Epub 2014 Jun 30. PMID 24980489
- [Background] Oberleithner H, Riethmuller C, Schillers H, MacGregor GA, de Wardener HE, Hausberg M. Plasma sodium stiffens vascular endothelium and reduces nitric oxide release. Proc Natl Acad Sci U S A. 2007 Oct 9;104(41):16281-6. doi: 10.1073/pnas.0707791104. Epub 2007 Oct 2. PMID 17911245
- [Background] Volpe M, Magri P, Rao MA, Cangianiello S, DeNicola L, Mele AF, Memoli B, Enea I, Rubattu S, Gigante B, Trimarco B, Epstein M, Condorelli M. Intrarenal determinants of sodium retention in mild heart failure: effects of angiotensin-converting enzyme inhibition. Hypertension. 1997 Aug;30(2 Pt 1):168-76. doi: 10.1161/01.hyp.30.2.168. PMID 9260976
- [Background] Nijst P, Verbrugge FH, Martens P, Dupont M, Tang WHW, Mullens W. Renal response to intravascular volume expansion in euvolemic heart failure patients with reduced ejection fraction: Mechanistic insights and clinical implications. Int J Cardiol. 2017 Sep 15;243:318-325. doi: 10.1016/j.ijcard.2017.05.041. Epub 2017 May 14. PMID 28545850
- [Background] McKie PM, Schirger JA, Costello-Boerrigter LC, Benike SL, Harstad LK, Bailey KR, Hodge DO, Redfield MM, Simari RD, Burnett JC Jr, Chen HH. Impaired natriuretic and renal endocrine response to acute volume expansion in pre-clinical systolic and diastolic dysfunction. J Am Coll Cardiol. 2011 Nov 8;58(20):2095-103. doi: 10.1016/j.jacc.2011.07.042. PMID 22051332
- [Background] Gaggin HK, Januzzi JL Jr. Biomarkers and diagnostics in heart failure. Biochim Biophys Acta. 2013 Dec;1832(12):2442-50. doi: 10.1016/j.bbadis.2012.12.014. Epub 2013 Jan 9. PMID 23313577
- [Background] Damman K, Van Veldhuisen DJ, Navis G, Vaidya VS, Smilde TD, Westenbrink BD, Bonventre JV, Voors AA, Hillege HL. Tubular damage in chronic systolic heart failure is associated with reduced survival independent of glomerular filtration rate. Heart. 2010 Aug;96(16):1297-302. doi: 10.1136/hrt.2010.194878. PMID 20659949